CLINICAL TRIAL: NCT06700304
Title: CAN-PRIME: An Early Feasibility Study of a Precise Robotically Implanted Brain-Computer Interface for the Control of External Devices
Brief Title: CAN-PRIME: Precise Robotically Implanted Brain-Computer Interface for the Control of External Devices
Acronym: CAN-PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuralink Corp (Industry)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N1-EFS-002
Record Dates: First submitted 2024-11-15; First posted 2024-11-21 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Tetraplegia/Tetraparesis; Quadriplegia; Quadriplegia/Tetraplegia; Cervical Spinal Cord Injury; Amyotrophic Lateral Sclerosis (ALS); Spinal Cord Injury (Quadraplegia); Spinal Cord Injury
Keywords: brain computer interface; Neuralink N1 Implant; Neuralink; Robot; tetraparesis; tetraplegia; quadriplegia; ALS; spinal cord injury; Amyotrophic lateral sclerosis; chip; brain chip; External device control; Wireless implant; Neuroprosthetics; SCI; paralysis
MeSH Terms: conditions — Quadriplegia; Amyotrophic Lateral Sclerosis; Spinal Cord Injuries; Paralysis

STUDY DESIGN:
Intervention Model Description: The study is a prospective, longitudinal, non-randomized, open-label, single-arm early feasibility study (EFS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAN-PRIME: Precise Robotically Implanted Brain-Computer Interface (Other): Open label
  Interventions: Device: N1 Implant; Device: R1 Robot

INTERVENTIONS:
Device: N1 Implant — The N1 Implant is a type of implantable brain-computer interface.
Device: R1 Robot — The R1 Robot is a robotic electrode thread inserter that implants the N1 Implant.

SUMMARY:
The CAN-PRIME Study is to test the safety and functionality of Neuralink's N1 Implant and R1 Robot in people who have difficulty moving their arms and legs (tetraparesis or tetraplegia). The N1 Implant is a small, wireless device placed in the skull. It connects to tiny threads inserted into the brain by the R1 Robot, which is a machine designed to carefully place these threads. This study will help researchers learn how well the implant and robot work and if they are safe for use.

ELIGIBILITY:
Inclusion Criteria:

* Severe quadriplegia (tetraplegia) due to spinal cord injury or amyotrophic lateral sclerosis (ALS) for at least 1 year without improvement, where quadriplegia is defined as having very limited or no hand, wrist, and arm movement and all levels below
* Life expectancy ≥ 12 months.
* Ability to communicate in English
* Presence of a stable caregiver

Exclusion Criteria:

* Moderate to high risk for serious perioperative adverse events
* Active implanted devices
* Morbid obesity (Body Mass Index > 40)
* History of poorly controlled seizures or epilepsy
* History of poorly controlled diabetes
* Requires magnetic resonance imaging (MRI) for any ongoing medical conditions
* Acquired or hereditary immunosuppression
* Use of smoking tobacco or other tobacco products
* Psychiatric or psychological disorder
* Brain MRI demonstrating hemorrhage, tumor, distorted or adverse anatomy.
* Any condition which, in the opinion of the Investigator, would compromise your ability to safely participate in the study or undergo the implantation procedure

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
The Rate of Device-Related Adverse Events (AE) | 12 months post-implant
The Rate of Procedure-Related Adverse Events (AE) | 12 months post-implant

SECONDARY OUTCOMES:
The Rate of Device-Related Adverse Events (AE) | Up to 36 months post-implant
The Rate of Procedure-Related Adverse Events (AE) | Up to 36 months post-implant
Change in Montreal Cognitive Assessment (MoCA) score during the Primary Study | From baseline to 3-, 6-, 9-, and 12-months post-implantation
Change in Montreal Cognitive Assessment (MoCA) score during the Long-term Follow-up Phase | From baseline to 36-months post-implantation
Change in Patient Health Questionnaire-9 (PHQ-9) score during the Primary Study | From baseline to 3-, 6-, 9-, and 12-months post-implantation
Change in Patient Health Questionnaire-9 (PHQ-9) score during the Long-term Follow-up Phase | From baseline to 36-months post-implantation
Change in Generalized Anxiety Disorder-7 (GAD-7) score during the Primary Study | From baseline to 3-, 6-, 9-, and 12-months post-implantation
Change in Generalized Anxiety Disorder-7 (GAD-7) score during the Long-term Follow-up Phase | From baseline to 36-months post-implantation

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuralink Website — https://neuralink.com/